CLINICAL TRIAL: NCT00002761
Title: CAMP-010: PHASE I/II STUDY OF IN VIVO PURGING FOLLOWED BY HIGH DOSE CHEMOTHERAPY, AUTOLOGOUS HEMATOPOIETIC STEM CELL INFUSION AND IMMUNOTHERAPY IN PATIENTS WITH CHRONIC MYELOID LEUKEMIA
Brief Title: Combination Chemotherapy Followed by Peripheral Stem Cell Transplantation in Treating Patients With Chronic Myelogenous Leukemia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Columbia University (Other)
Purpose: Treatment
Other Study IDs: AAAA7158; CU-CAMP-10; NCI-V96-0873
Record Dates: First submitted 1999-11-01; First posted 2003-11-24 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Leukemia
Keywords: relapsing chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; chronic myelogenous leukemia, BCR-ABL1 positive
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Filgrastim; Interferon-gamma; Busulfan; Cyclophosphamide; Cyclosporine; Cytarabine; Idarubicin; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Biological: recombinant interferon gamma
Drug: busulfan
Drug: cyclophosphamide
Drug: cyclosporine
Drug: cytarabine
Drug: idarubicin
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase I/II trial to study the effectiveness of combination chemotherapy followed by peripheral stem cell transplantation in treating patients with chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether intensive idarubicin and cytarabine leads to adequate harvest of Philadelphia chromosome-negative peripheral blood stem cells (PBSC) in patients with chronic myelogenous leukemia in chronic phase. II. Determine the toxicity of this intensive regimen in these patients. III. Determine the graft-versus-leukemia effect induced in these patients by cyclosporine and interferon gamma post-PBSC transplantation. IV. Determine the transformation-free and overall survival in patients treated with a high-dose conditioning regimen comprising busulfan and cyclophosphamide followed by PBSC transplantation plus immunotherapy.

OUTLINE: Patients receive idarubicin IV and cytarabine IV over 2 hours on days 1-3. When blood counts recover, Philadelphia chromosome negative peripheral blood stem cells (PBSC) are harvested. Filgrastim (G-CSF) is administered subcutaneously (SC) beginning 24 hours after completion of cytarabine infusion and continuing until blood counts have recovered for 3 consecutive days after harvest of PBSC. Patients with more than 5% blasts in marrow or any peripheral blasts, interferon resistance, interferon intolerance with poor prognosis, and clonal evolution proceed to conditioning followed by PBSC transplantation. Patients receive conditioning comprising oral busulfan every 6 hrs on days -8 to -5 and cyclophosphamide IV over 2 hours on days -4 and -3. PBSC are reinfused on day 0. Patients receive graft versus leukemia induction comprising cyclosporine IV over 4 hours every 12 hours on days 0-28 and interferon gamma SC beginning on day 7 and continuing every other day through day 28. Patients are followed every 3 months for 1 year and then annually for 5 years.

PROJECTED ACCRUAL: A total of 15-43 patients will be accrued for this study within 4-8 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of chronic myelogenous leukemia in first chronic phase Philadelphia chromosome-positive Myelofibrosis less than 3+ on bone marrow biopsy Ineligible for allogeneic transplantation No suitable allogeneic sibling donor OR Under 55 years old but refuses unrelated donor transplantation or no unrelated donor available

PATIENT CHARACTERISTICS: Age: 18 to physiologic 60 Performance status: ECOG 0-1 Hematopoietic: See Disease Characteristics WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 2 times normal (unless elevation due to Gilbert's disease) SGOT less than 1.5 times normal Renal: Creatinine less than 1.5 times normal Cardiovascular: Left ventricular ejection fraction at least 50% Pulmonary: DLCO at least 60% predicted Other: HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior interferon alfa Chemotherapy: No concurrent conventional chemotherapy Endocrine therapy: No concurrent steroids during chemotherapy Radiotherapy: Not specified Surgery: Not specified Other: No concurrent barbiturates or acetaminophen during chemotherapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 1996-02; Primary Completion 2007-02 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gwen L. Nichols, MD, Study Chair — Herbert Irving Comprehensive Cancer Center

REFERENCES:
- [Background] Papadopoulos KP, Nichols G: Autologous peripheral blood progenitor (PBPC) transplantation in patients with chronic myeloid leukemia. Biol Blood Marrow Transplant 4(2): A-55, 109, 1998.